CLINICAL TRIAL: NCT02747043
Title: A Randomized, Double-Blind Study Evaluating the Efficacy, Safety and Immunogenicity of ABP 798 Compared With Rituximab in Subjects With CD20 Positive B-Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Study to Assess if ABP798 is Safe & Effective in Treating Non Hodgkin Lymphoma Compared to Rituximab
Acronym: JASMINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130109; 2013-005542-11 (EudraCT Number)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: CD20 Positive B-cell Non-Hodgkin Lymphoma; ABP 798
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABP 798 (Experimental): ABP 798 was administered at a dose of 375 mg/m^2 as an intravenous (IV) infusion once weekly for 4 weeks followed by dosing at weeks 12 and 20.
  Interventions: Biological: ABP 798
- Rituximab (Active Comparator): Rituximab was administered at a dose of 375 mg/m^2 as an IV infusion once weekly for 4 weeks followed by dosing at weeks 12 and 20.
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: ABP 798 — ABP 798 was supplied as a sterile, preservative-free liquid concentrate for IV infusion at a concentration of 10 mg/mL in either 100 mg/10 mL or 500 mg/50 mL single-dose vials. Subjects were to receive premedications before each infusion. Premedications were to be given according to local practice for administration of rituximab therapy.
  Other Names: biosimilar to rituximab
  Arms: ABP 798
Biological: Rituximab — Rituximab was procured from commercial supplies in the US and was supplied as a sterile, clear, colorless, preservative-free liquid concentrate for IV infusion at a concentration of 10 mg/mL in either 100-mg/10 mL or 500-mg/50 mL single-dose vials. Subjects were to receive premedications before each infusion. Premedications were to be given according to local practice for administration of rituximab therapy.
  Other Names: Rituxan
  Arms: Rituximab

SUMMARY:
This was a randomized, double-blind, active-controlled, multiple-dose, clinical similarity study to evaluate the efficacy, pharmacokinetics, pharmacodynamics, safety, tolerability and immunogenicity of ABP 798 compared with rituximab in subjects with grade 1, 2, or 3a follicular B-cell NHL and low tumor burden.

Subjects were randomized in a 1:1 ratio to receive a 375 mg/m^2 intravenous infusion of either ABP 798 or rituximab once weekly for 4 weeks followed by dosing at weeks 12 and 20.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older
* Histological confirmed (by lymph node or extranodal region biopsy), Grade 1, 2, or 3a follicular B-cell NHL expressing CD20 within 12 months before randomization
* Stage 2, 3, or 4 (per Cotswold's Modification of Ann Arbor Staging System) with measurable disease (per International Working Group)

  * subjects must have a baseline scan (computed tomography [CT]) of the neck (if palpable lymph node > 1.0 cm), chest, abdomen, and pelvis to assess disease burden within 6 weeks before randomization
  * subjects must have had a baseline bone marrow biopsy within 12 months before randomization. Previously confirmed positive bone marrow involvement does not need to be repeated for purposes of screening.
* Low tumor burden based on the Groupe d'Etudes des Lymphomes Folliculaires (GELF) criteria

  * largest nodal or extranodal mass ≤ 7 cm
  * no more than 3 nodal sites with diameter > 3 cm
  * no splenomegaly > 16cm by CT scan and no symptomatic splenomegaly
  * no significant pleural or peritoneal serous effusions by CT
  * lactate dehydrogenase ≤ upper limit of normal (ULN)
  * no B symptoms (night sweats, fever [temperature > 38°C], weight loss > 10% in the previous 6 months)

Exclusion Criteria:

* Diffuse large cell component and/or Grade 3b follicular NHL
* History or known presence of central nervous system metastases
* Malignancy other than NHL within 5 years (except treated in-situ cervical cancer, or squamous or basal cell carcinoma of the skin)
* Recent infection requiring a course of systemic anti-infective agents that was completed ≤ 7 days before randomization (with the exception of uncomplicated urinary tract infection)
* Other investigational procedures that can impact the study data, results, or patient safety while participating in this study are excluded; participation in observational studies is allowed.
* Subject is currently enrolled in or has not yet completed at least 30 days or 5 half-lives (whichever is longer) since ending other investigational device or drug study(s), including vaccines, or subject is receiving other investigational agent(s)
* Previous use of either commercially available or investigational chemotherapy, biological, or immunological therapy for NHL (including rituximab or biosimilar rituximab, or other anti-CD20 treatments)
* Systemic corticosteroid use within 3 months before randomization (inhaled are allowable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (88):
- United States (5):
  - Research Site, Encinitas, California
  - Research Site, Mount Sterling, Kentucky
  - Research Site, Billings, Montana
  - Research Site, Zanesville, Ohio
  - Research Site, Roanoke, Virginia
- Australia (3):
  - Research Site, Gosford, New South Wales
  - Research Site, Frankston, Victoria
  - Research Site, Perth, Western Australia
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Stara Zagora
- Research Site, Windsor, Ontario, Canada
- Colombia (2):
  - Research Site, Medellín, Antioquia
  - Research Site, Bogota, Cundinamarca
- Czechia (2):
  - Research Site, Prague, Prague
  - Research Site, Ostrava - Poruba, Severomoravsky KRAJ
- France (6):
  - Research Site, Bordeaux, Aquitaine
  - Research Site, Clermont-Ferrand, Auvergne
  - Research Site, Cesson-Sévigné, Brittany Region
  - Research Site, Boulogne-sur-Mer, Hauts-de-France
  - Research Site, La Rochelle, Poitou-charentes
  - Research Site, Poitiers, Poitou-charentes
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Germany (7):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Augsburg, Bavaria
  - Research Site, Würzburg, Bavaria
  - Research Site, Kassel, Hesse
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Leipzig, Saxony
  - Research Site, Flensburg, Schleswig-Holstein
- Greece (2):
  - Research Site, Athens, Attica
  - Research Site, Patra, Peloponnese
- India (7):
  - Research Site, Surat, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Bikaner, Rajasthan
- Research Site, Be’er Ya‘aqov, Rehoboth, Israel
- Italy (12):
  - Research Site, San Giovanni Rotondo, Foggia
  - Research Site, Bergamo, Lombardy
  - Research Site, Pesaro, Pesaro E Urbino
  - Research Site, Aviano, Pordenone
  - Research Site, Candiolo, Torino
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, Terni
- Japan (8):
  - Research Site, Chiba, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Kobe, Hyōgo
  - Research Site, Tsu, Mie-ken
  - Research Site, Utsunomiya, Tochigi
  - Research Site, Tachikawa, Tokyo
  - Research Site, Tokyo
- Mexico (2):
  - Research Site, Mexico City, Mexico City
  - Research Site, Chihuahua City
- Poland (4):
  - Research Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Legnica, Lower Silesian Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
- Romania (3):
  - Research Site, Târgu Mureş, Mureș County
  - Research Site, Timișoara, Timiș County
  - Research Site, Bucharest
- South Korea (6):
  - Research Site, Seoul, Gyeonggi-do
  - Research Site, Jinju, Gyeongsangnam-do
  - Research Site, Pusan, Gyeongsangnam-do
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Ulsan
- Spain (9):
  - Research Site, Sabadell, Barcelona
  - Research Site, Córdoba, Cordoba
  - Research Site, Majadahonda, Madrid
  - Research Site, La Laguna Tenerife, Santa CRUZ DE Tenerife
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Cáceres
  - Research Site, Madrid
  - Research Site, Salamanca
- Ukraine (4):
  - Research Site, Kyiv, Kyiv City
  - Research Site, Uzhhorod, Zakarpattia Oblast
  - Research Site, Chernivtsi
  - Research Site, Dnipropetrovsk

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Niederwieser D, Hamm C, Cobb P, Mo M, Forsyth C, Tucci A, Hanes V, Delwail V, Hajek R, Chien D. Efficacy and Safety of ABP 798: Results from the JASMINE Trial in Patients with Follicular Lymphoma in Comparison with Rituximab Reference Product. Target Oncol. 2020 Oct;15(5):599-611. doi: 10.1007/s11523-020-00748-4. PMID 33044684
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 380 subjects were screened and 256 participants (128 in the ABP 798 treatment group and 128 in the rituximab treatment group) were randomized at 91 centers across 20 countries.
Pre-assignment Details: Participants were randomized centrally to receive either ABP 798 or rituximab in a 1:1 manner. The randomization was stratified based on geographic region (Europe, Americas, Japan, Asia Pacific - Other) and age group (> 60 years of age, ≤ 60 years of age).
Period: Overall Study
Arm/Group | ABP 798 | Rituximab
Started | 128 | 128
Treated | 128 | 126
Completed (Completed Week 28) | 118 | 123
Not Completed | 10 | 5
Not completed — Other | 1 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Disease progression | 4 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 798 | Rituximab | Total
Number analyzed (Participants) | 128 | 128 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.72) | 58.2 (12.20) | 57.9 (12.45)
Age, Customized [Count of Participants; unit: Participants]
  <= 60 years | 71 | 70 | 141
  > 60 years | 57 | 58 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 62 | 130
  Male | 60 | 66 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 102 | 101 | 203
  Asian, Non-Japanese | 17 | 14 | 31
  Asian, Japanese | 7 | 8 | 15
  Missing | 1 | 2 | 3
  Other | 0 | 2 | 2
  American Indian or Alaska Native | 1 | 0 | 1
  White, Asian-Non-Japanese | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 119 | 119 | 238
  Hispanic or Latino | 8 | 7 | 15
  Not allowed to collect | 1 | 2 | 3
Weight [Mean (Standard Deviation); unit: kg] | 75.29 (19.135) | 75.19 (16.981) | 75.24 (18.063)
Height [Mean (Standard Deviation); unit: cm] | 166.81 (10.737) | 167.64 (10.292) | 167.22 (10.506)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0 | 107 | 110 | 217
    Grade 1 | 21 | 18 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 88 | 86 | 174
  Asia Pacific - Other | 23 | 23 | 46
  Americas | 10 | 11 | 21
  Japan | 7 | 8 | 15
Time Since Original Diagnosis [Mean (Standard Deviation); unit: months] | 6.31 (16.325) | 5.17 (10.181) | 5.74 (13.590)
Previous Radiation Treatment [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 6
  No | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Responded (Overall Response Rate - ORR) by Week 28 Based on Independent Central Assessment of Disease
Description: Overall response within the first treatment cycle was assessed according to International Working Group - Non-Hodgkin Lymphoma criteria (IWG-NHL criteria [Cheson et al, 1999]) by a central reader. Response was evaluated using computerized tomography (CT) scans and positron emission tomography (PET) (to assess nodal disease/organ enlargement), and bone marrow biopsy (to assess bone marrow infiltration). ORR was the percentage of participants with a best overall response of complete response (CR), unconfirmed complete response (CRu) or partial response (PR). Participants that do not meet the criteria for response were considered non-responders.
  CR was defined as no evidence of disease. CRu showed nodes in the original sum of the products (SPD) regressed by >75% and/or indeterminate bone marrow results.
  PR was a ≥ 50% decrease in SPD of the six largest dominant nodes; >=50% decrease in liver and spleen nodes, and no increase in size of other nodes nor any new sites of disease.
Time Frame: Post treatment up to Week 28
Population: The modified full analysis set included all randomized participants with evidence of disease at baseline per the tumor assessment from the central, independent, blinded assessments. Analyses for the modified full analysis set was based on randomized treatment assignment.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 123 | 124
percentage of participants | 78.0 [70.7 to 85.4] | 70.2 [62.1 to 78.2]
Statistical Analysis 1: Comparison: ABP 798 vs Rituximab; Test type: Equivalence — Clinical equivalence of the primary endpoint will first be demonstrated by comparing the 1-sided 95% lower confidence limit of the RD of ORR by week 28 between ABP 798 and rituximab with a noninferiority margin of -15%. If this is successful, the 1-sided upper 95% confidence limit of the RD of ORR by week 28 will be compared with a nonsuperiority margin of +35.5%; Risk Difference (RD) = 7.7, 90% CI 2-sided [-1.4 to 16.8] — The 2-sided 90% confidence limits of the risk difference (RD) of ORR by week 28 used a generalized linear model adjusted for the stratification factors (geographic region and age group)
Statistical Analysis 2: Comparison: ABP 798 vs Rituximab; Test type: Other; Risk Difference (RD) = 7.7, 95% CI 2-sided [-3.2 to 18.6]

2. Secondary Outcome: Percentage of Participants Who Responded (Overall Response Rate - ORR) at Week 12 Based on Independent Central Assessment of Disease
Description: as for outcome 1
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 123 | 124
percentage of participants | 59.3 [50.7 to 68.0] | 58.1 [49.4 to 66.7]
Statistical Analysis 1: Comparison: ABP 798 vs Rituximab; The 2-sided 90% confidence limits of the risk difference (RD) of ORR at week 12 used a generalized linear model adjusted for the stratification factors (geographic region and age group); Test type: Other; Risk Difference (RD) = 0.9, 90% CI 2-sided [-9.3 to 11.2]
Statistical Analysis 2: Comparison: ABP 798 vs Rituximab; The 2-sided 95% confidence limits of the risk difference (RD) of ORR at week 12 used a generalized linear model adjusted for the stratification factors (geographic region and age group); Test type: Other; Risk Difference (RD) = 0.9, 95% CI 2-sided [-11.3 to 13.2]

3. Secondary Outcome: Pharmacokinetic Serum Concentrations by Visit
Description: Pharmacokinetic serum samples were analyzed by a central lab. Lower limit of quantification (LLOQ) was 0.25 ug/mL. PK concentrations below the lower limit of quantification were assigned a value of 0. Geometric mean and geometric CV were only calculated using concentrations >0.
Time Frame: Weeks 2, 3, 4, 12 and 20
Population: Safety Analysis Set of participants with available data. Participants with PK concentrations below the lower limit of quantification (LLOQ) were excluded from these analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 126
microgram/mL
  Week 2 (predose): number analyzed (Participants) | 123 | 125
  Week 2 (predose) | 58.66 (50.4) | 58.63 (76.9)
  Week 3 (predose): number analyzed (Participants) | 125 | 126
  Week 3 (predose) | 105.39 (37.8) | 108.77 (59.1)
  Week 4 (predose): number analyzed (Participants) | 126 | 121
  Week 4 (predose) | 132.70 (42.6) | 140.23 (57.9)
  Week 12 (predose): number analyzed (Participants) | 121 | 124
  Week 12 (predose) | 21.86 (156.1) | 20.55 (194.1)
  Week 12 (postdose): number analyzed (Participants) | 113 | 117
  Week 12 (postdose) | 207.05 (58.1) | 209.14 (66.8)
  Week 20 (predose): number analyzed (Participants) | 118 | 122
  Week 20 (predose) | 13.37 (138.7) | 16.45 (115.8)

4. Secondary Outcome: Percentage of Participants With Complete Depletion of Clusters of Differentiation 19-Positive (CD19+) Cell Count From Baseline to Day 8
Description: Complete depletion of CD19+ cell count at any postdose time was defined as CD19+ cell counts < 20 cell/μL (0.02 * 10^9 cell/L). Participants with missing CD19+ cell count at baseline or participants with CD19+ cell count < 20 cell/μL at baseline were to be excluded from the derivation of complete depletion of CD19+ cell count.
Time Frame: Baseline (Day 1), Study Day 8
Population: Full analysis set of participants with available data. Participants with missing CD19+ cell count at baseline or participants with CD19+ cell count < 20 cell/μL at baseline were to be excluded from the derivation of complete depletion of CD19+ cell count.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 115 | 116
percentage of participants | 98.3 | 98.3

5. Secondary Outcome: Total Immunoglobulin G (IgG) Results by Visit
Description: Samples were analyzed by a central lab.
Time Frame: Baseline (Day 1), Day 8 (Week 2), Weeks 3, 4, 28
Population: Full analysis set of participants with available data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 128
g/L
  Baseline: number analyzed (Participants) | 127 | 123
  Baseline | 9.740 (2.5988) | 10.570 (2.5970)
  Day 8 (Week 2): number analyzed (Participants) | 122 | 123
  Day 8 (Week 2) | 9.790 (2.5719) | 10.486 (2.4916)
  Week 3: number analyzed (Participants) | 122 | 123
  Week 3 | 9.545 (2.5933) | 10.374 (2.3214)
  Week 4: number analyzed (Participants) | 124 | 121
  Week 4 | 9.744 (2.5805) | 10.196 (2.2842)
  Week 28: number analyzed (Participants) | 103 | 104
  Week 28 | 9.846 (2.6316) | 10.281 (2.3617)

6. Secondary Outcome: Total Immunoglobulin M (IgM) Results by Visit
Description: Samples were analyzed by a central lab.
Time Frame: Baseline (Day 1), Day 8 (Week 2), Weeks 3, 4, 28
Population: Full analysis set of participants with available data.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 128
g/L
  Baseline: number analyzed (Participants) | 127 | 123
  Baseline | 1.021 (1.0072) | 1.247 (3.4018)
  Day 8 (Week 2): number analyzed (Participants) | 122 | 123
  Day 8 (Week 2) | 1.004 (1.0300) | 1.280 (3.7292)
  Week 3: number analyzed (Participants) | 122 | 122
  Week 3 | 1.001 (1.0564) | 1.370 (5.0250)
  Week 4: number analyzed (Participants) | 124 | 120
  Week 4 | 0.985 (1.0459) | 1.385 (5.3266)
  Week 28: number analyzed (Participants) | 103 | 104
  Week 28 | 0.816 (0.8505) | 1.127 (3.6752)

7. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment. Each AE was graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, where Grade 1 = Mild AE Grade 2 = Moderate AE Grade 3 = Severe AE Grade 4 = Life-threatening or disabling AE Grade 5 = Death related to AE. Serious adverse events include any event that is fatal, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or other significant medical hazard.
  IP = investigational product
Time Frame: Day 1 (post treatment) to Week 28
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 126
Participants
  Any AE | 107 | 95
  Any grade >=3 AE | 14 | 13
  Any fatal AE | 0 | 0
  Any serious AE | 5 | 5
  Any AE leading to discontinuation of IP | 4 | 1
  Any AE leading to dose delay/withheld IP | 9 | 9

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events of Interest (AEOIs)
Description: The AEOIs prespecified for this study were infusion reactions including hypersensitivity, cardiac disorders, serious infections, progressive multifocal leukoencephalopathy, hematological reactions, hepatitis B reactivation, opportunistic infections, severe mucocutaneous reactions, tumor lysis syndrome, gastrointestinal perforation, and reversible posterior leukoencephalopathy syndrome.
  Infusion reactions including hypersensitivity adverse events of interest must have start date the same as, or one day after, an investigational product administration start date.
Time Frame: Day 1 (post treatment) to Week 28
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 126
percentage of participants
  Any AEOI | 49.2 | 45.2
  Infusion reactions including hypersensitivity | 43.0 | 42.9
  Hematological reactions | 5.5 | 4.8
  Cardiac disorders | 2.3 | 1.6
  Serious infections | 1.6 | 0
  Severe mucocutaneous reactions | 0.8 | 0
  Gastrointestinal perforation | 0 | 0
  Hepatitis B reactivation | 0 | 0
  Opportunistic infection | 0 | 0
  Progressive multifocal leukoencephalopathy | 0 | 0
  Reversible posterior leukoencephalopathy | 0 | 0
  Tumor lysis syndrome | 0 | 0
Statistical Analysis 1: Comparison: ABP 798 vs Rituximab; Percentage risk difference for 'Any adverse event of interest'; Test type: Other — Risk difference (ABP 798 - Rituximab) and CIs were estimated by Wald asymptotic confidence limits, or exact confidence limits if n < 25 for either treatment; Risk Difference (RD) = 4.0, 95% CI 2-sided [-8.3 to 16.3]
Statistical Analysis 2: Comparison: ABP 798 vs Rituximab; Percentage risk difference for 'Infusion reactions including hypersensitivity'; Test type: Other — [test comment as in outcome 8, analysis 1]; Risk Difference (RD) = 0.1, 95% CI 2-sided [-12.1 to 12.3]
Statistical Analysis 3: Comparison: ABP 798 vs Rituximab; Percentage risk difference for 'Hematological reactions'; Test type: Other — [test comment as in outcome 8, analysis 1]; Risk Difference (RD) = 0.7, 95% CI 2-sided [-11.8 to 13.0]
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab; Percentage risk difference in 'Cardiac disorders'; Test type: Other — [test comment as in outcome 8, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-11.8 to 13.2]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab; Percentage risk difference in 'Serious infections'; Test type: Other — [test comment as in outcome 8, analysis 1]; Risk Difference (RD) = 1.6, 95% CI 2-sided [-10.9 to 14.0]
Statistical Analysis 6: Comparison: ABP 798 vs Rituximab; Percentage risk difference in 'Severe mucocutaneous reactions'; Test type: Other — [test comment as in outcome 8, analysis 1]; Risk Difference (RD) = 0.8, 95% CI 2-sided [-11.7 to 13.2]

9. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies
Description: Samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect antibodies capable of binding to ABP 798/rituximab (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based assay to determine neutralizing activity against ABP 798/rituximab (Neutralizing Antibody Assay).
  Developing antibody incidence was defined as participants with a negative or no binding antibody result at baseline and a positive antibody result at any post-baseline time point.
Time Frame: Baseline (Day 1), Weeks 12, 20 and 28
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 126 | 123
Participants
  Binding antibody positive | 3 | 1
  Neutralizing antibody positive | 1 | 1

10. Secondary Outcome: Participants' Progression-Free Survival (PFS) Status Based on the Independent Central Assessment of Disease
Description: PFS was based on disease assessments determined by the central, independent, blinded radiologists' and oncologist's review.
Time Frame: Day 1 up to Week 28
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 126
percentage of participants
  Participants with disease progression or death | 3.1 | 2.4
  Participants alive and progression-free | 96.9 | 97.6

11. Secondary Outcome: Percentage of Participants Who Survived -- Overall Survival (OS)
Description: Percentage of participants who were alive at the end of the study.
Time Frame: Day 1 up to Week 28
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab
Number analyzed (Participants) | 128 | 126
percentage of participants | 100 | 100

ADVERSE EVENTS:
Time Frame: Day 1 to 28 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | ABP 798 | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/126
Serious Adverse Events (participants affected / at risk) | 5/128 | 5/126
Other Adverse Events (participants affected / at risk) | 59/128 | 61/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 798 (N=128) | Rituximab (N=126)
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 798 (N=128) | Rituximab (N=126)
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 9
Nausea (Gastrointestinal disorders) | 6 | 14
Asthenia (General disorders) | 12 | 6
Fatigue (General disorders) | 13 | 12
Pyrexia (General disorders) | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 1
Headache (Nervous system disorders) | 15 | 12
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 12
Rash (Skin and subcutaneous tissue disorders) | 9 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02747043/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT02747043/SAP_001.pdf